CLINICAL TRIAL: NCT05053321
Title: Reduction of Demoralization in Patients With Tardive Dyskinesia After Treatment With Valbenazine
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funding.
Sponsor: Yale University (Other)
Collaborators: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000031423; No NIH funding (Other: 11.09.23)
Record Dates: First submitted 2021-09-13; First posted 2021-09-22 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Tardive Dyskinesia
MeSH Terms: conditions — Tardive Dyskinesia | interventions — valbenazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Valbenazine (Experimental): All participants will be treated with Valbenazine for 6 weeks.
  Interventions: Drug: Valbenazine

INTERVENTIONS:
Drug: Valbenazine — All participants will be treated with Valbenazine for 6 weeks.

SUMMARY:
This will be an Investigator-initiated pilot study in which participants will be assessed with various scales to measure demoralization, anxiety, depression, and subjective incompetence at baseline and every two weeks after treatment with Valbenazine for a total of 6 weeks. Improvement in TD will be assessed as well and correlated with reduction in demoralization.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 26-84
2. Sex: Both males and females will be included
3. Diagnosis of dopamine receptor-blocker induced tardive dyskinesia according to the DSM-5 criteria: "involuntary athetoid or choreiform movements lasting at least a few weeks, developing in association with the use of a neuroleptic medication for at least a few months, and persisting beyond 4-8 weeks"

Exclusion Criteria:

The following classes of patients will be excluded:

1. Patients with unstable psychiatric status defined as having a total score on BPRS of 50 or higher
2. Patients who have suicidal or homicidal ideation, intent, or plan or viewed as having a significant risk of suicidal or violent behavior;
3. Patients with cognitive impairment as defined by a score of 24 or less on the MMSE
4. Patients with current diagnosis of alcohol or substance use disorder made according to DSM-5 criteria
5. Patients with clinically significant unstable medical condition defined as follows: a comorbid abnormal movement disorder more prominent than tardive dyskinesia (e.g., parkinsonism, akathisia, truncal dystonia), a score of greater than 2 on two or more items of the Simpson-Angus Scale, or a history of neuroleptic malignant syndrome.
6. Patients previously treated with Valbenazine or any other medication specifically indicated for tardive dyskinesia
7. Patients currently taking strong CYP3A4 inducers, dopamine agonists, MAO inhibitors, stimulants, and/or VMAT2 inhibitors
8. Patients with congenital long QT syndrome or arrhythmias associated with prolonged QT interval
9. Patients with risk factors for prolonged QT such as electrolyte abnormalities (hypokalemia, hypocalcemia, hypomagnesemia), anorexia nervosa, diuretic use, certain heart conditions, and other medical conditions
10. Patients tested positive for Coronavirus Covid-19
11. Patients with impaired decision-making capacity
12. Institutionalized individuals
13. Prisoners

Ages: 26 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-18 (Actual); Primary Completion 2025-10-18 (Estimated); Study Completion 2025-10-18 (Estimated)

PRIMARY OUTCOMES:
Change in demoralization Scale | Baseline, week 2, week 4, and week 6
  The change in symptoms of demoralization will be measured using the Demoralization Scale-II (DS-II). Scale scores range from 0 (minimum) to 32 (maximum), with higher scores indicating more demoralization (i.e., a worse outcome). Reduction of score to below 10 will be measured

SECONDARY OUTCOMES:
Change in subjective incompetence scale (SIS) score | Baseline, week 2, week 4, and week 6
  The SIS consists of 12 items, each item has 4 response alternatives scored as 0, 1, 2, 3. The scores range from 0 to 36. Higher scores mean more severe subjective incompetence.

CONTACTS AND LOCATIONS:
Overall Officials: John De Figueiredo, MD, Principal Investigator — Clinical Professor of Psychiatry
Locations (1):
- Yale Church Street Research Unit., New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared after a reasonable request and after the project is completed. It will be shared with the sponsor and deposited .